CLINICAL TRIAL: NCT00350116
Title: Topical Vitamin B12 in Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1-Stucker
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2006-07-10 (Estimated); Status verified 2006-07

CONDITIONS: Chronic Plaque Psoriasis
Keywords: plaque psoriasis; Vitamin B12
MeSH Terms: interventions — Vitamin B 12

INTERVENTIONS:
Drug: topical vitamin B12

SUMMARY:
Objective: To test the efficacy and tolerability of a vitamin B12 cream for the treatment of chronic plaque psoriasis.

Design: Multicenter, double-blind, randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
Objective: To test the efficacy and tolerability of a vitamin B12 cream for the treatment of chronic plaque psoriasis.

Design: Multicenter, double-blind, randomized, placebo-controlled trial. Setting: ambulatory patients in research or referral centers. Patients: Volunteer sample of 51 patients with chronic plaque psoriasis. Interventions: All Patients applied vitamin B12 cream twice daily for 8 weeks to one side of the body and placebo to the other.

Main outcome measures: Modified Psoriasis Area and Severity Index (PASI) at weeks 0, 2, 4, 6 and 8. Thickness and density of 3 references plaques determined by 20 MHz sonography. Assessment of efficiency and tolerability by patients and investigators.

ELIGIBILITY:
Inclusion Criteria:

* 18years
* chronic plaque psoriasis

Exclusion Criteria:

* incapability of Vitamin B12
* necessity of systemic therapy
* use of other potentially psoriasis modifying drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2001-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Main outcome measures: Modified Psoriasis Area and Severity Index (PASI) at weeks 0, 2, 4, 6 and 8. Thickness and density of 3 references plaques determined by 20 MHz sonography. Assessment of efficiency and tolerability by patients and investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Altmeyer, Prof. Dr., Principal Investigator — Ruhr University Bochum, Dep. Dermatology and Allergology
Locations (1):
- Dep. Dermatology and Allergology, Ruhr-University Bochum, Bochum, Germany